CLINICAL TRIAL: NCT05390320
Title: Dental and Periodontal Changes Following the Acceleration of Decrowding of Lower Anterior Teeth Using a PAOO Procedure: A Randomized Controlled Trial
Brief Title: Dental and Periodontal Changes Following the Acceleration of Alignment of Crowded Lower Anterior Teeth Using a Surgical Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-10-2022
Record Dates: First submitted 2022-05-20; First posted 2022-05-25 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Crowding, Tooth
Keywords: PAOO; moderate crowding; gingival index; plaque index; papillary bleeding index
MeSH Terms: conditions — Malocclusion | interventions — Orthodontic Appliances, Fixed

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Periodontally accelerated osteogenic orthodontics (Experimental): The patients in this group will be treated by periodontally accelerated osteogenic orthodontics using fixed appliances.
  Interventions: Procedure: PAOO
- Conventional treatment (Active Comparator): The patients in this group will be treated using fixed appliances and conventional treatment without any surgical intervention to accelerate tooth movement.
  Interventions: Other: Fixed appliance

INTERVENTIONS:
Procedure: PAOO — Periodontally accelerated osteogenic orthodontics will be applied to treat patients with moderate crowding.
  Arms: Periodontally accelerated osteogenic orthodontics
Other: Fixed appliance — Fixed appliances will be applied to treat patients with moderate crowding without any acceleration methods.
  Arms: Conventional treatment

SUMMARY:
Patients at the Orthodontic Department of the University of Damascus Dental School will be examined and subjects who meet the inclusion criteria will be included. Then, initial diagnostic records (diagnostic gypsum models, internal and external oral photographs, and radiographic images) will be studied to ensure that the selection criteria are accurately matched.

This study aims to compare two groups of patients with moderate crowding of the lower anterior teeth. Experimental group: the patients in this group will be treated with periodontally accelerated osteogenic orthodontics Control group: the patients in this group will be treated using fixed appliances without any acceleration method.

DETAILED DESCRIPTION:
Correction of irregular teeth can take a long time, and this depends on various factors such as the good compliance of the patient, the amount of dental crowding, and the need for extraction in the course of orthodontic treatment.

Many methods have been used to accelerate tooth movement, and recently the PAOO technique has emerged as an effective therapeutic intervention.

PAOO is a promising procedure but only a few cases were reported in the literature. Controlled clinical and histological studies are needed to understand the biology of tooth movement with this procedure, the effect on teeth and bone, post-retention stability, measuring the volume of mature bone formation, and determining the status of the periodontium and roots after treatment.

ELIGIBILITY:
Inclusion Criteria:

* skeletal class I malocclusion (ANB=2-4)
* normal vertical growth pattern.
* moderate crowding of lower anterior teeth (i.e., 4-6 millimeters of a tooth size-arch length discrepancy)
* 1 to 3 mm of overjet and 1 to 4 mm of the overbite
* good oral health

Exclusion Criteria:

* medical, social, and psycho contraindications to oral surgery
* presence of periodontal diseases
* poor oral hygiene
* previous orthodontic treatment

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-10-06 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Change in Little's Index of Irregularity | T0: one day before the beginning of treatment; T1: after 1 month; T2: after 2 months; T3: after 4 months; T4: after 5 months; T5: at the end of the alignment stage which is expected within 5 - 6 months
  The irregularity of the lower incisors is calculated by measuring the amount of deviations of the anatomic contact points between the six anterior teeth in the horizontal direction in mm, since the sum of these measurements represents the value of the index (Little, 1975).
  The ordinary orthodontic treatment aims to keep this Index less than 1 mm at the end of treatment.
Change in the inter-canine width | T0: One day before the beginning of treatment; T1: at the end of the alignment stage
  The distance between the cusp tips of the lower canines. This variable will be measured on plaster models.
Change in the inter-2nd premolar width | T0: One day before the beginning of treatment; T1: at the end of the alignment stage
  The distance between the central fossae of the lower second premolars. This variable will be measured on plaster models.

SECONDARY OUTCOMES:
Change in the Gingival index | T0: One day before the beginning of treatment; T1: at the end of the alignment stage
  Measured by degrees at each tooth: (0) Normal gingival; (1) mild inflammation; (2) Moderate inflammation; (3) severe inflammation
Change in the Plaque index | T0: One day before the beginning of treatment; T1: at the end of the alignment stage
  Measured by degrees at each tooth: (0) No plaque; (1) thin plaque layer; (2) moderate plaque layer; (3) severe plaque along the gingival margin
Change in the Papillary Bleeding Index | T0: One day before the beginning of treatment; T1: at the end of the alignment stage
  Measured by the severity of any bleeding: (0) No bleeding; (1) a single discreet bleeding point; (2) several isolated bleeding points; (3) the interdental triangle fills with blood shortly after probing; (4) profuse bleeding occurs after probing.

CONTACTS AND LOCATIONS:
Overall Officials: Hallaj I Alsino, DDS, Principal Investigator — Department of orthodontics, Damascus University, Syria; Mohammad Y Hajeer, DDS,MSc,PhD, Study Director — Department of orthodontics, Damascus University, Syria; Issam Khoury, DDS,MSc,PhD, Study Director — Department of Oral and Maxillofacial Surgery, Damascus University, Syria
Locations (1):
- University of Damascus, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yu H, Jiao F, Wang B, Shen SG. Piezoelectric decortication applied in periodontally accelerated osteogenic orthodontics. J Craniofac Surg. 2013;24(5):1750-2. doi: 10.1097/SCS.0b013e3182902c5a. PMID 24036771
- [Background] Wu J, Jiang JH, Xu L, Liang C, Bai Y, Zou W. A pilot clinical study of Class III surgical patients facilitated by improved accelerated osteogenic orthodontic treatments. Angle Orthod. 2015 Jul;85(4):616-24. doi: 10.2319/032414-220.1. Epub 2014 Oct 27. PMID 25347045
- [Background] Bahammam MA. Effectiveness of bovine-derived xenograft versus bioactive glass with periodontally accelerated osteogenic orthodontics in adults: a randomized, controlled clinical trial. BMC Oral Health. 2016 Nov 30;16(1):126. doi: 10.1186/s12903-016-0321-x. PMID 27903250
- [Background] Amit G, Jps K, Pankaj B, Suchinder S, Parul B. Periodontally accelerated osteogenic orthodontics (PAOO) - a review. J Clin Exp Dent. 2012 Dec 1;4(5):e292-6. doi: 10.4317/jced.50822. eCollection 2012 Dec 1. PMID 24455038
- [Background] Nowzari H, Yorita FK, Chang HC. Periodontally accelerated osteogenic orthodontics combined with autogenous bone grafting. Compend Contin Educ Dent. 2008 May;29(4):200-6; quiz 207, 218. PMID 18533317